CLINICAL TRIAL: NCT03903146
Title: Early Childhood Obesity Risk Reduction Program in Hispanics
Brief Title: Childhood Risk Reduction Program in Hispanics
Acronym: ECOR-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Maria Linares (Other)
Responsible Party: Sponsor-Investigator, Ana Maria Linares, Associate Professor of Nursing, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-0164-P2H
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Breast Feeding, Exclusive
Keywords: Breastfeeding; Exclusive breastfeeding; Hispanic Women; Kentucky
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to intervention or control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: To decrease the feeling of discomfort if the mother was not breastfeeding her infant, the trained research staff collecting data on infant feeding status at T-4, T-5, and T-6 remain blinded to the participant's group. To assure that the research staff remain blinded a script was created that explained the importance that the participant abstained to share with research staff if she was getting the visit of any other research personnel. The script was consistently read to participants in each encounter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group of participants was assigned to receive the intervention by the bicultural/bilingual team of Peer counselor and Lactation Consultant. An intensive support intervention (1 prenatal visit, 1 in-hospital visit, 1 home postpartum visit, and free phone calls) were conducted individually to mothers participating until 6 months after the birth of the infant.
  Interventions: Behavioral: Early Childhood Obesity Risk-Reduction Program in Hispanics
- Control Group (No Intervention): All participants in this group received traditional prenatal care in the clinic and received the usual educational material (in their proficient language) about breastfeeding during prenatal care provided by the Special Supplemental Nutritional for Women, Infants, and Children (WIC) program implemented in the clinics. Women were also able to receive one breastfeeding consultation during their hospital stay in the birthing center as part of the actual protocol established in the UK Chandler Hospital (Baby-friendly Hospital that includes support of breastfeeding during hospital stay). Women in the usual care group did not have any contact with the study IBCLC/PC.

INTERVENTIONS:
Behavioral: Early Childhood Obesity Risk-Reduction Program in Hispanics — Sessions Prenatal (40 min): Includes a colorful binder with information about breastfeeding. Set her goals and action plan for breastfeeding. Past experiences with breastfeeding. Benefits of adopting a healthy behavior, describe and discuss infant feeding and qualms about mixed feeding, barriers to EBF and self-efficacy.
  Prenatal Calls (10 min.): Discuss strategies available to accomplish mother's breastfeeding goals. Answer questions. Follow-up call until delivery.
  Hospital visit (30 min.): PC visit mother at the hospital stay to support the participant in her effort to breastfeeding.
  Postpartum home-visit (40 min.) IBCLC performs a home visit to assess infant feeding pattern, breastfeeding techniques with hands-on assistance if needed. Provide supplemental breastfeeding devices as needed. Answer all questions.
  Postpartum calls (10 min.): PC/IBCLC ask about problems/concerns and answer questions. Repeat phone calls as needed (at least 1 a month).
  Other Names: Promoting Exclusive breastfeeding in Hispanic Mothers
  Arms: Intervention Group

SUMMARY:
Childhood obesity is a serious problem in the United States, as it increases the risk for various cardiometabolic, pulmonary, and psychosocial complications for children, which often continue into adulthood. Examination of disparities in early childhood obesity among ethnic groups shows that Hispanic infants/children have higher rates of overweight and obesity than children/infants of other races/ethnicities. According to the most recent National Health and Nutrition Examination Survey (2014), the prevalence of high weight for recumbent length (≥95th percentile) among infant and toddlers from birth to 2 years was 6.6% in Whites, 8.4% in Blacks, and 9.4% in Hispanics. Furthermore, the percentages of children ages 2 through 5 years who are overweight or obese (Body Mass Index [BMI] ≥ 85th) were 20.9% among non-Hispanic Whites, 21.9% among non-Hispanic Blacks, and 29.8% among Hispanics. These data suggest that ethnic disparities in childhood obesity prevalence have their origins in the earliest stages of life.

Bergmann et al. reported that infants that received early formula artificial feeding by 3 months had significantly higher BMIs and thicker skin fold than exclusively breastfed infants, and from 6 months on, compared with breastfed children, a consistently higher proportion of artificially-fed children exceeded the 90th and 97th percentile of BMI and skin folder thickness reference values. Exclusive breastfeeding (EBF), defined as exclusive infant feeding with breast milk without any additional food or drink, is the feeding option engendering greatest nutrition and health, imparting enhanced glucose management and reductions in early childhood obesity.

Hispanic mothers in the U.S. are more likely to supplement with formula in the first 2 days of life, compared with Black and White U.S. mothers (Hispanic 33%; Black 28%; White 22%). Additionally, a common feeding practice among Hispanic mothers is the early introduction of solids including ethnic food. The introduction of formula or complementary food in breastfed Hispanic infants produces an overfeeding problem that leads to childhood obesity. In a study published by this team of investigators on infant feeding management in Hispanic women living in Kentucky was reported that even when 51% of the group of Hispanic mothers initiated EBF during hospital stay, only 22% continued EBF at 4 months after birth. These trends underscore the critical need for intervention to support EBF in this population.

Objectives: There is great opportunity and immense need to empower vulnerable, at-risk Hispanic mother/infant dyads to prevent and manage childhood obesity by increasing duration and EBF and delaying the introduction of complementary food. The primary aim of this pilot study was to determinate the feasibility and evaluate the clinical impact of a novel, tailored, culturally and linguistically appropriate community-based intervention. The intervention was delivered by Hispanics bilingual/bicultural team of an International Board Certified Lactation Consultant (IBCLC) and a peer counselor (PC) and was tested in terms of its influence on key modifiable factors that are positively associated with increasing breastfeeding duration and exclusivity: (a) mother's breastfeeding intention; (b) breastfeeding self-efficacy; and (c) perceived social support. Specific aims for this study are:

Aim 1: Determine the feasibility of the intervention. This aim is designed to answer the following important research questions:

Q-1: Is the planned recruitment period sufficient to enroll the targeted number of participants? Q-2: What percent of treatment group participants will complete all sessions of the intervention? Q-3: What percent of participants will be retained in the study until the conclusion? Q-4: What factors are associated with intervention adherence and study retention?

Aim 2: Evaluate the clinical impact of the intervention. The following hypotheses will be tested:

Hypothesis #1: Women in the intervention group will have higher intention to breastfeed during the pre-natal period and will perceive greater self-efficacy and social support during postnatal period, compared with the usual care group.

Hypothesis #2: Women in the intervention group will be more likely to initiate EBF during their post-delivery in-hospital stay than those in the usual care group.

Hypothesis #3: Among those who practice EBF during their hospital stay, women in the intervention group will be more likely to continue EBF for six months than women in the usual care group.

Hypothesis #4: Women in the intervention group will have longer time to introduction of complementary food to their infants compared with the usual care group.

DETAILED DESCRIPTION:
The feasibility of a tailored community-based intervention, entitled Early Childhood Obesity Risk-Reduction Program in Hispanics (ECOR-H), was tested. The ECOR-H provided mothers with culturally tailored, self-management risk-reduction modules, and with continued peer counselor (PC) and professional lactation consultant support to develop personal skill-set to "take control" of modifiable behaviors and help participants to exclusively breastfeed for a longer time and delay the introduction of solid food to the infants. The study was conducted in the University of Kentucky (UK) Polk Dalton Clinic and in the Birthing Center of UK Albert B. Chandler Hospital. A convenient sample of 39 self-identified Hispanic pregnant women were recruited and randomly assigned to intervention and standard care groups (Intervention n = 20 ; Control n=19).

Trained Research Personnel (RP) approached and screened women for eligibility in the waiting prenatal area, which was exclusively used by pregnant women--while waiting for prenatal care appointments. Screening for eligibility was accomplished using a checklist that contains eligibility criteria. If the woman satisfied the eligibility criteria, the potential participant was invited to go to a private room in the clinic available for this purpose and the research staff provided a review and explanation of the study with an invitation to participate. If the person stated that was not interested, the research staff asked if can share the reason(s) why of the decision and collected the information in the log track of potential recruitment contacted. Then the research staff thanked the time and ended the conversation. Women who agreed to participate were scheduled for an appointment at another convenient time at the participant's home or clinic to provide informed consent and signed a HIPAA authorization. Since the potential participants included English/Spanish speaking participants, the informed consent, HIPPA authorization, and interview materials and intervention sessions were provided in the language in which the subject was most proficient. The parental permission for the infant was included in the informed consent that the mother signed when agreed to participate in the study. The consent form explains that this study would collect information on the infant from the medical record. The type of information that would be collected about the infant was also described in the HIPAA authorization form. The informed consent form provided the overall goal of the research; a brief description of the research; the type of survey that would be conducted in each encounter; the infant assessment for the anthropometric measurements of weight, length, and head circumference, and the mother's BMI. The explanation also described the minimal risks to participants and the potential benefits, procedures to assure confidentiality, and the voluntary nature of participation and how the confidentiality of the information that participants provide during the study would be maintained. It was also necessary to collect the name and a telephone number for contact information and follow-up encounters. The research staff explained that this information would be used only for research purposes and to send reminding of time, date, and place of the follow-up interviews, and it will be destroyed by the end of the study.

All identifiers such as name, address, date of birth, telephone number, medical record number, and a code number were included in a private list and saved in a Microsoft Excel program with password protection to which only the PI and research staff had access. The Microsoft Excel file was opened only in encrypted computers located in the office of the PI and research staff in the University of Kentucky College of Nursing. Only staff certified in human subjects research and who were listed as study personnel with the University of Kentucky Institutional Review Board (UK IRB) were allowed access to participant data. When the study was completed, the data was de-identified prior to data sharing.

After providing informed consent, the participant completed a baseline study survey. Following the baseline interview, the research staff informed the PI weekly of the new number of participants recruited. The PI randomly assigned participants to intervention and standard care groups following randomization procedures. Data collection was similar for both groups (standard care and intervention) and was obtained independently by research staff at 30 weeks of pregnancy (T-1), at 37 or more weeks of pregnancy (T-2), chart review of mother/infant medical record at birth (T-3), between 2-4 weeks after birth (T-4), and at three (T-5) and six (T-6) months after the birth. Randomization: After the baseline interview (T-1), the participant was randomly assigned to the standard of care group or standard care plus ECOR-H intervention group. The random assignment schedule was stratified according to whether the woman was a first-time mother or has other children; this allowed equal numbers within each of these two strata to be assigned to each of the two treatment conditions. The biostatistician prepared envelopes that contain the treatment assignments, one set for each stratum. Within each stratum, the treatment assignments were set in blocks of 10 (i.e., 5 assignments to each of the treatment conditions). Though the total recruitment target was 39 women, it was not known what percentage will be first-time mothers, so the investigators created at least 3 blocks of 10 mothers for each of the two strata. The blocks in the randomization schedule ensured that investigators have approximately equivalent numbers of mothers in each of the treatment and standard care groups at all stages of data collection for both strata. The PI opened the sealed envelope based in the parity of the participant; each envelope contained a card with "Standard care" or "Intervention." The PI informed the PC the participants that have been assigned to initiate the intervention. The PC initiated contact with the participant in a time frame not longer than a week. The research personnel who collected data was blinded to the treatment condition of the participants. A script was read in each data collection session to request the participant to avoid sharing with the research staff if she was or not receiving the visit of the PC or professional lactation consultant.

Data Analysis: Given the descriptive nature of this feasibility study, no power analysis was warranted. However, the feasibility study informed effect sizes that will be used to estimate statistical power for future studies, including a planned R01 submission. Descriptive analysis will be accomplished using means and standard deviations or frequency distributions. Differences in baseline demographic and personal characteristics between the intervention and usual care groups will be assessed using two-sample t-tests, Mann-Whitney U tests, or chi-square tests of association to verify that the randomization yielded comparable groups from this population. Measures of feasibility (including number of participants completing the intervention sessions and entire study) will be examined. Logistic regression with demographics and personal characteristics as covariates will be used to discern whether there is a difference in the likelihood of breastfeeding initiation, duration and exclusivity between the intervention and usual care group. Qualitative methods will be used to assess factors impacting recruitment, adherence, and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Immigrant Hispanic women;
* pregnant at or beyond 30 weeks of gestation;
* intention to at least try to breastfeed;
* planning to deliver at a local birthing hospital; and
* planning to remain in Central Kentucky for at least 6 months after the birth of their child.

Exclusion Criteria:

* prior or current participation in any study to enhance breastfeeding;
* pregnant with twins;
* history of breast surgery;
* contraindication to BF (e.g., HIV-positive status, chronic therapy with medications incompatible with BF, alcohol dependence or other substance abuse); and
* presumed or known congenital fetus defects.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurnani M, Birken C, Hamilton J. Childhood Obesity: Causes, Consequences, and Management. Pediatr Clin North Am. 2015 Aug;62(4):821-40. doi: 10.1016/j.pcl.2015.04.001. Epub 2015 May 23. PMID 26210619
- [Background] Kelishadi R, Farajian S. The protective effects of breastfeeding on chronic non-communicable diseases in adulthood: A review of evidence. Adv Biomed Res. 2014 Jan 9;3:3. doi: 10.4103/2277-9175.124629. eCollection 2014. PMID 24600594
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Bergmann KE, Bergmann RL, Von Kries R, Bohm O, Richter R, Dudenhausen JW, Wahn U. Early determinants of childhood overweight and adiposity in a birth cohort study: role of breast-feeding. Int J Obes Relat Metab Disord. 2003 Feb;27(2):162-72. doi: 10.1038/sj.ijo.802200. PMID 12586995
- [Background] Palou A, Sanchez J, Pico C. Nutrient-gene interactions in early life programming: leptin in breast milk prevents obesity later on in life. Adv Exp Med Biol. 2009;646:95-104. doi: 10.1007/978-1-4020-9173-5_10. PMID 19536667
- [Background] Spatz DL. Preventing obesity starts with breastfeeding. J Perinat Neonatal Nurs. 2014 Jan-Mar;28(1):41-50. doi: 10.1097/JPN.0000000000000009. PMID 24476651
- [Background] Centers for Disease Control and Prevention C. Final Formula Supplementation of Breast Milk Rates by Socio-demographic Factors, Among Children Born in 2006. 2012c; http://www.cdc.gov/breastfeeding/data/NIS_data/2006/socio-demographic_formula.htm, 2012.
- [Background] Cartagena DC, Ameringer SW, McGrath J, Jallo N, Masho SW, Myers BJ. Factors contributing to infant overfeeding with Hispanic mothers. J Obstet Gynecol Neonatal Nurs. 2014 Mar-Apr;43(2):139-59. doi: 10.1111/1552-6909.12279. Epub 2014 Feb 6. PMID 24502196
- [Background] Wright AL, Holberg C, Taussig LM. Infant-feeding practices among middle-class Anglos and Hispanics. Pediatrics. 1988 Sep;82(3 Pt 2):496-503. PMID 3405686
- [Background] Gill SL. Breastfeeding by Hispanic women. J Obstet Gynecol Neonatal Nurs. 2009 Mar-Apr;38(2):244-52. doi: 10.1111/j.1552-6909.2009.01013.x. PMID 19323721
- [Background] Linares AM, Rayens MK, Dozier A, Wiggins A, Dignan MB. Factors influencing exclusive breastfeeding at 4 months postpartum in a sample of urban Hispanic mothers in Kentucky. J Hum Lact. 2015 May;31(2):307-14. doi: 10.1177/0890334414565711. Epub 2015 Jan 16. PMID 25596411
- [Background] Thulier D. A call for clarity in infant breast and bottle-feeding definitions for research. J Obstet Gynecol Neonatal Nurs. 2010 Nov-Dec;39(6):627-34. doi: 10.1111/j.1552-6909.2010.01197.x. PMID 21044147
- [Background] Nommsen-Rivers LA, Cohen RJ, Chantry CJ, Dewey KG. The Infant Feeding Intentions scale demonstrates construct validity and comparability in quantifying maternal breastfeeding intentions across multiple ethnic groups. Matern Child Nutr. 2010 Jul 1;6(3):220-7. doi: 10.1111/j.1740-8709.2009.00213.x. PMID 20929494
- [Background] Linares AM, Hall L, Ashford K. Psychometric Testing of the Autonomy and Relatedness Inventory-Spanish Version. J Nurs Meas. 2015;23(1):E27-37. doi: 10.1891/1061-3749.23.1.E27. PMID 26269139
- [Background] Wambach KA, Aaronson L, Breedlove G, Domian EW, Rojjanasrirat W, Yeh HW. A randomized controlled trial of breastfeeding support and education for adolescent mothers. West J Nurs Res. 2011 Jun;33(4):486-505. doi: 10.1177/0193945910380408. Epub 2010 Sep 27. PMID 20876551
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Marin G, Sabogal F, Marin BV, Otero-Sabogal R, Perez-Stable EJ. Development of a Short Acculturation Scale for Hispanics. Hispanic Journal of Behavioral Sciences. 1987;9 (2 ):183-205
- [Background] Meedya S, Fahy K, Kable A. Factors that positively influence breastfeeding duration to 6 months: a literature review. Women Birth. 2010 Dec;23(4):135-45. doi: 10.1016/j.wombi.2010.02.002. Epub 2010 Mar 17. PMID 20299299
- [Result] 13th Breastfeeding and Feminism International Conference: The Dance of Nurture in a Complex World: How Biology, Gender, and Social Context Shape How We Nourish Our Children. J Hum Lact. 2018 Aug;34(3):600-630. doi: 10.1177/0890334418776646. Epub 2018 Jun 21. No abstract available. PMID 29928830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 06.23.2016 and ended 03.31.2017 N=40 participants. Recruited in an outpatient clinic, Prenatal care area.
Groups:
- Intervention Group: This group of participants was assigned to receive the intervention by the bicultural/bilingual team of Peer counselor and Lactation Consultant. An intensive support intervention (1 prenatal visit, 1 in-hospital visit, 1 home postpartum visit, and free phone calls) were conducted individually to mothers participating until 6 months after the birth of the infant.
  Early Childhood Obesity Risk-Reduction Program in Hispanics: Sessions Prenatal (40 min): Includes a colorful binder with information about breastfeeding. Set her goals and action plan for breastfeeding. Past experiences with breastfeeding. Benefits of adopting a healthy behavior, describe and discuss infant feeding and qualms about mixed feeding, barriers to EBF and self-efficacy.
  Prenatal Calls (10 min.): Discuss strategies available to accomplish mother's breastfeeding goals. Answer questions. Follow-up call until delivery.
  Hospital visit (30 min.): PC visit mother at the hospital stay to support the participant in her effort to breastfeeding.
  Postpartum home-visit (40 min.) IBCLC performs a home visit to assess infant feeding pattern, breastfeeding techniques with hands-on assistance if needed. Provide supplemental breastfeeding devices as needed. Answer all questions.
  Postpartum calls (10 min.): PC/IBCLC ask about problems/concerns and answer questions. Repeat phone calls as needed (at least 1 a month).
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 20 | 20
Completed (At least completed 80% of the intervention modules.) | 14 | 15
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (1.15) | 26.5 (1.51) | 25.4 (.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanics | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breastfeeding (EBF)
Description: Infant Feeding Status was determined at discharge via medical chart review from reports in the infant's chart. Follow-up infant feeding status at each encounter post-discharge, was assessed via mother's report; mothers were asked to choose the practice that most closely resembles how she was feeding her infant with possible options of exclusive breastfeeding, predominant breast milk; mixed feeding; predominant formula milk; and exclusive formula milk. Then, the mother was also asked 'Does your baby receive water, juice or any other juices or solids?' If the mother agreed that the infant is receiving additional food, mothers were asked when they introduced the food to their child and portions given by day.
Time Frame: At hospital discharge
Population: 1 participant withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
Participants
  EBF at Discharge | 9 | 4
  Breastfeeding supplementing with formula | 11 | 13
  Only formula feeding | 0 | 2

2. Secondary Outcome: Intention to Breastfeed
Description: Infant Feeding Intention was assessed at baseline and again before the birth of the infant using the Infant Feeding Intentions Scale, Spanish version (IFI). This scale has 5 items, with response options ranging from 0 = 'Very much disagree' to 4 = 'Very much agree.' The total score is obtained by averaging the first 2 items (which include planning about giving breastfeeding a try and another item that is reverse-coded as it is an endorsement of planning to use formula) and adding the remaining 3 items to this mean. The range of scores is from 0 to 16, with higher scores indicating a stronger intention to EBF for 6 months. Cronbach's alpha for this sample was 0.87.
Time Frame: Prenatal: At baseline (around 30 weeks of pregnancy) and after 37 week of pregnancy.
Population: Number of participants differ due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale
  Baseline (30 weeks) | 13.0 (6.4) | 10.3 (5.2)
  37 weeks: number analyzed (Participants) | 16 | 12
  37 weeks | 14.37 (1.92) | 10.33 (5.3)

3. Secondary Outcome: Social Support
Description: Social support was assessed during the prenatal period using the Spanish version of the Autonomy and Relatedness Inventory (ARI). Each of the 32 items is scored on a 5-point scale, with response options ranging from 1 = 'Not at all like' to 5 = 'Very much like.' To calculate a total score, negative items are reversed, all ratings are summed, and then 32 is subtracted from the sum so that the cumulative score ranges from 0 to 128. Higher scores indicate a more positive assessment of the relationship.
Time Frame: prenatal at baseline
Population: 5 participants did not complete questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 17 | 18
score on a scale | 120.76 (1.98) | 121.67 (2.68)

4. Secondary Outcome: Knowledge of Breastfeeding
Description: Breast Feeding (BF) Knowledge was assessed at baseline and again before the birth of the infant using an adapted Spanish version of the BF Knowledge Questionnaire. The questionnaire has 25 items, with response options 1= True, and 0 = False. The total score is obtained by first reversing eight of the items by assigning a value of 1 for each correct answer of 'False' and then adding all the items. The range of scores is from 0 to 25, with higher scores indicating a greater knowledge of BF. Kuder-Richardson 20 for this sample was 0.72.
Time Frame: Prenatal: At baseline (around 30 weeks of pregnancy) and after 37 weeks of pregnancy.
Population: Number of Participants differ due to attrition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale
  Baseline (30 weeks) | 20.1 (3.1) | 18.8 (3.9)
  37 weeks: number analyzed (Participants) | 16 | 16
  37 weeks | 21.75 (3.0) | 19.0 (3.38)

5. Secondary Outcome: Breastfeeding Self-Efficacy
Description: Breastfeeding Self-Efficacy Scale-Short Version (BSES) was used to measure maternal confidence to breastfeed during postpartum. This instrument consists of 14 items, each with a response set ranging from 1 = 'Not at all confident' to 5= 'Very confident.' The summary score is created by adding the 14 items in the scale, with scores ranging from 14 to 70; higher scores indicated greater self-efficacy for breastfeeding.
Time Frame: Post natal at 1, 3, 6 months postpartum only when woman was breastfeeding.
Population: Breastfeeding Self-efficacy (BFSE) at 1 month (n=30), and 3 months (n=19), and 6 months after birth (n=16). These numbers reflect participants that were still breastfeeding. These numbers do not include formula only participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
score on a scale
  BFSE at 1 month after Delivery | 60.06 (2.54) | 62.28 (1.76)
  BFSE at 3 months: number analyzed (Participants) | 11 | 8
  BFSE at 3 months | 65.0 (9.25) | 64 (4.2)
  BFSE at 6 months: number analyzed (Participants) | 9 | 7
  BFSE at 6 months | 66 (2.35) | 61.29 (1.88)

6. Other Pre Specified Outcome: Acculturation
Description: The 7-item short version of the Hispanic Acculturation Scale assessed the likelihood of using Spanish or English in different situations. Responses are rated in a five-point choice: only Spanish; Spanish better than English; both equally; English better than Spanish; and only English. The responses are summed, with the total score ranging from 5 to 35, with higher scores indicating a greater degree of acculturation.
Time Frame: At Baseline around 30 weeks of pregnancy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
units on a scale | 13 (1.9) | 10.3 (5.2)

7. Primary Outcome: Exclusive Breastfeeding (EBF)
Description: as for outcome 1
Time Frame: 3 months
Population: (N=34), participants lost to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 17 | 17
Participants
  EBF | 7 | 2
  Breastfeeding supplementing with formula | 4 | 6
  Only formula feeding | 6 | 9

8. Primary Outcome: Exclusive Breastfeeding (EBF)
Description: as for outcome 1
Time Frame: 6 months
Population: (N=29), participants lost to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 15
Participants
  EBF | 7 | 1
  Breastfeeding supplementing with formula | 2 | 6
  Only formula feeding | 5 | 8

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03903146/Prot_SAP_001.pdf